CLINICAL TRIAL: NCT06244303
Title: Clinical Research Study to Assess the Efficacy of Two Brushing Regimens: 1) a Toothpaste Containing Stannous Fluoride With a Mouthwash Containing Cetylpyridinium Chloride and a Manual Toothbrush as Compared to 2) a Regular Fluoride Toothpaste and Standard Manual Toothbrush in the Reduction of Established Dental Plaque and Gingivitis.
Brief Title: Clinical Research Study to Assess the Efficacy of Two Brushing Regimens in the Reduction of Established Dental Plaque and Gingivitis.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRO-2023-11-PG-DWN-CA-BGS
Record Dates: First submitted 2024-01-29; First posted 2024-02-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-01

CONDITIONS: Gingivitis; Plaque
Keywords: Loe and Silness Gingival Index; Quigley and Hein Plaque Index
MeSH Terms: conditions — Gingivitis; Plaque, Amyloid

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group I (Active Comparator): manual Tooth Brush + Colgate Total TP (0.454% SnF, 1100 ppm F) Brush 2 x day / 2 mins Colgate Total Mouthwash (CPC+Zn) Swish 20 mL / 30 secs
  Interventions: Drug: manual Tooth Brush + Colgate Total TP (0.454% SnF, 1100 ppm F); Drug: manual toothbrush + Colgate dental cream
- Group II (Placebo Comparator): Manual Toothbrush +Colgate Great Regular Flavor Toothpaste Brush w/ full ribbon, 2x day / 2mins
  Interventions: Drug: manual Tooth Brush + Colgate Total TP (0.454% SnF, 1100 ppm F); Drug: manual toothbrush + Colgate dental cream

INTERVENTIONS:
Drug: manual Tooth Brush + Colgate Total TP (0.454% SnF, 1100 ppm F) — Toothpaste, toothbrush & mouthwash regime
Drug: manual toothbrush + Colgate dental cream — toothpaste + toothbrush

SUMMARY:
Qualified subjects will be enrolled and randomized to one of the two study groups based on their initial Plaque and Gingivitis scores. Subjects will be instructed to use the products according to the instructions provided. Subjects will return to the dental office for evaluation after 1-, 3-, 6-, and 12-weeks of unsupervised product use at home. All subjects will be followed for adverse events throughout the study

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form.
* Male and female subjects aged 18-70 years, inclusive.
* Availability for the twelve-week duration of the clinical research study.
* Good general health based on the opinion of the study investigator
* Minimum of 20 permanent natural teeth (excluding third molars).
* Initial gingivitis index of at least 1.0 as determined by the use of the Loe and Silness Gingival Index.
* Initial plaque index of at least 1.5 as determined by the use of the Quigley and Hein Plaque Index (Turesky Modification)

Exclusion Criteria:

* Presence of orthodontic appliances.
* Presence of partial removable dentures.
* Tumor(s) of the soft or hard tissues of the oral cavity.
* Moderate and/or advanced periodontal disease, rampant caries, or any condition that the dental examiner considers exclusionary from the study.
* Five or more carious lesions requiring immediate restorative treatment.
* Antibiotic use any time during the one-month period prior to entry into the study.
* Participation in any other clinical study or test panel within the one month prior to entry into the study.
* Dental prophylaxis during the past two weeks prior to baseline examinations.
* History of allergies to oral care/personal care consumer products or their ingredients.
* On any prescription medicines that might interfere with the study outcome.
* An existing medical condition that prohibits eating and/or drinking for periods up to 4 hours.
* History of alcohol and/or drug abuse.
* Self-reported pregnancy and/or lactating subjects

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2024-01-22 (Actual); Primary Completion 2024-04-16 (Estimated); Study Completion 2024-04-16 (Estimated)

PRIMARY OUTCOMES:
Quigley and Hein Plaque Index | Baseline, 1-, 3-, 6-, and 12-week
  reductions in dental plaque
Loe and Silness Gingival Index | Baseline, 1-, 3-, 6-, and 12-week
  reductions in gingivitis

CONTACTS AND LOCATIONS:
Overall Officials: Farid Ayad, B.D.S., D.D.S., MSC, Principal Investigator — FAR Oral and Systemic Health Consulting, Inc
Locations (1):
- Mesa Dental Centre, Costa Mesa, California, United States

IPD SHARING:
Plan to Share IPD: No